CLINICAL TRIAL: NCT06929013
Title: Monitoring of Blood Clearance Kinetics of the Nucleosome and CTCF in Peri-operative Management of Peritoneal Metastasis Colorectal Cancer.
Brief Title: Blood Clearance Kinetics of the Nucleosome and CTCF in Peritoneal Metastasis Colorectal Cancer.
Acronym: NUCLEAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_0852
Record Dates: First submitted 2025-03-25; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Peritoneal Carcinomatosis; Peritoneal Metastases From Colorectal Cancer
Keywords: Biomarkers; Peritoneal carcinomatosis; CTCF; Nucleosome
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective multicohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Peritoneal metastases colorectal cancer (Experimental): * Peritoneal metastases colorectal cancer histologically proven
  * Synchronous or metachronous peritoneal metastases.
  * Patients eligible for initial cytoreduction surgery.
  * Non mucinous tumor (mucinous cells contingent <30%).
  Interventions: Biological: Blood sampling
- Colorectal cancer (Experimental): Histologically proven colorectal cancer with no known metastatic
  Interventions: Biological: Blood sampling
- Non-oncological chronic inflammatory diseases (Experimental): Surgery for inflammatory bowel disease (Crohn's, chronic ulcerative colitis) such as ileocaecal resection, colectomy, and bowel resection.
  Interventions: Biological: Blood sampling
- Non-malignant diseases (Experimental): Non-inflammatory and non-oncological diseases:
  * Parietal repairs.
  * Elective sigmoidectomy for diverticulosis
  Interventions: Biological: Blood sampling
- Abdominal sepsis conditions (Experimental): * Peritonitis due to digestive perforation in non-oncological pathology.
  * Non-perforated appendicitis.
  * Cholecystitis.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Inclusion (baseline): 28 mL Incision (surgery): 18 mL End surgery: 18 mL H+12 after end surgery: 18 mL H+4 after end surgery: 18 mL H+48 after end surgery: 18 mL H+72 after end surgery: 18 mL D+7 after end surgery: 18 mL D+14 after surgery: 18 mL 4 to 6 weeks after surgery:28 mL

SUMMARY:
Colorectal cancer is highly prevalent in France, ranking second among women and third among men. Its primary metastatic sites include the liver, lungs, and peritoneum. For peritoneal metastases, when the disease is moderately extensive, cytoreductive surgery is recommended in an expert centre. Following this procedure, the surgeon uses the CC-Score (Completeness of Cytoreduction after Surgery Score) to assess the completeness of surgical resection by evaluating the largest remaining tumor residue. This subjective score is currently the main prognostic factor for oncological outcomes post-surgery. However, there is no objective score based on biological criteria to evaluate the radicality of resection, despite the hypothesis that the micrometastatic component of the disease could be biologically assessed using appropriate circulating markers.

New biomarkers are emerging and appear relevant for determining the presence of tumor residual disease. Notable among these are circulating tumor DNA, which can detect mutated DNA released by tumor cells into the patient's blood through high-throughput sequencing, and new markers related to epigenetic modifications in cancer cells. These markers target specific nucleosomes or the transcription factor CTCF and show promise in detecting residual disease.

To effectively use these markers for constructing a biological score to detect residual disease in peritoneal carcinomatosis, it is essential to understand their perioperative kinetics. This is crucial because cellular debris release is expected post-surgery, necessitating the determination of the most relevant time point for measurement. Additionally, these markers appear to be correlated with blood inflammation levels, requiring a description of this correlation to account for this potential confounding factor. Finally, the sensitivity and specificity of these markers must be determined by studying their perioperative kinetics in patient groups undergoing surgeries other than cytoreductions for peritoneal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Common criteria:

  * Male/female over 18 years of age.
  * Weight ≥ 55 kg at inclusion.
  * Signature of a free and informed consent form.
* Specific criteria:

Group 1:

* Peritoneal metastases colorectal cancer histologically proven
* Synchronous or metachronous peritoneal metastases.
* Patients eligible for initial cytoreduction surgery.
* Non mucinous tumor (mucinous cells contingent <30%).

Group 2:

Colorectal cancer

Group 3:

Non-oncological chronic inflammatory diseases

Group 4:

Non-oncological chronic inflammatory diseases : parietal repairs, elective sigmoidectomy for diverticulosis

Group 5:

Abdominal sepsis conditions: peritonitis due to digestive perforation in non-oncological pathology, non-perforated appendicitis, cholecystitis.

Non inclusion Criteria:

* Patient with an active cancer (excluding colorectal cancer).
* Person with a progressive autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Kinetic of nucleosome and CCCTC-binding factor (CTCF) | From the inclusion (baseline) to 4 to 6 weeks after surgical procedure.
  Blood clearance kinetics of the nucleosome (H3K27me3, H3K36me3, H3.1 et H3K9me3) and CCCTC-binding factor (CTCF).

SECONDARY OUTCOMES:
Kinetic of inflammatory markers - Albumin | From the inclusion (baseline) to 4 to 6 weeks after surgical procedure.
  Blood clearance kinetics of albumin
Kinetic of inflammatory markers - C-reactive protein | From the inclusion (baseline) to 4 to 6 weeks after surgical procedure.
  Blood clearance kinetics of C-reactive protein
Kinetic of inflammatory markers - Interleukin IL-6 | From the inclusion (baseline) to 4 to 6 weeks after surgical procedure.
  Blood clearance kinetics of Interleukin IL-6
Correlation between inflammatory markers, nucleosome and CCCTC-binding factor (CTCF). | Completed postoperative follow-up : at least 4 to 6 weeks after surgery
  Correlation test between blood concentration of inflammatory markers (albumin, C-reactive protein, Interleukin IL-6), nucleosome nucleosome (H3K27me3, H3K36me3, H3.1 et H3K9me3) and CCCTC-binding factor (CTCF).
Nucleosome and CCCTC-binding factor (CTCF) sensitivity and specificity | Completed postoperative follow-up : at least 4 to 6 weeks after surgery
  To assess the sensitivity and specificity of the nucleosome and CCCTC-binding factor (CTCF) blood clearance kinetic for the colorectal cancer peritoneal metastatic condition

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France